CLINICAL TRIAL: NCT01035593
Title: Recombinant Human C1 Inhibitor for the Treatment of Early Antibody-Mediated Rejection in Renal Transplantation
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Recent improvements in clinical practice have reduced the apparent incidence of AMR in renal transplantation.
Sponsor: Pharming Technologies B.V. (Industry)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C1 2201
Record Dates: First submitted 2009-12-16; First posted 2009-12-18 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Graft Rejection; Kidney Transplantation
MeSH Terms: interventions — Plasmapheresis; Immunoglobulins, Intravenous; conestat alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (PP + IVIG) (Active Comparator): Plasmapheresis and IVIG 100mg/kg every other day x 5 treatments
  Interventions: Procedure: plasmapheresis and IVIG
- PP + IVIG + rhC1INH (Experimental): Plasmapheresis + 100mg/kg IVIG every other day x 5 treatments plus rhC1Inh 100u/kg IV daily x 7 consecutive days (once daily on PP days, twice daily on non-PP days).
  Interventions: Drug: recombinant C1 inhibitor

INTERVENTIONS:
Procedure: plasmapheresis and IVIG — Plasmapheresis with either 5% human albumin or FFP replacement, plus IVIG 100mg/kg IV after each PP session, every other day x 5 treatments
  Arms: Standard of Care (PP + IVIG)
Drug: recombinant C1 inhibitor — 100units/kg IV for seven consecutive days (once daily on PP/IVIG days, twice daily on non-PP/IVIG days).
  Arms: PP + IVIG + rhC1INH

SUMMARY:
The purpose of this study will be to assess the safety, tolerability, and efficacy of rhC1INH in renal transplant recipients with biopsy-confirmed antibody-mediated rejection (AMR) within 30 days of renal transplantation. This study will combine the investigational drug rhC1INH with a standard regimen of plasmapheresis (PP) and intravenous immune globulin (IVIG) and compare this to PP and IVIG alone.

DETAILED DESCRIPTION:
This is an Investigator-initiated, prospective, open-label, randomized, adaptive design study to enroll 30 adult renal transplant recipients with biopsy-confirmed AMR within 30 days post transplantation. After informed consent is obtained and study eligibility is confirmed, subjects will be enrolled immediately after biopsy confirmation of AMR and positive donor specific antibody (DSA). Subjects will then be randomized into one of two treatment groups (SOC [control] or rhC1INH). An initial cohort of 8 subjects (3 SOC, 5 rhC1INH) will receive intensive safety monitoring of the coagulation system and for thromboembolic events.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of renal transplantation within 30 days prior to enrollment.
* AMR documented by light microscopic changes and immunohistochemical C4d staining on renal biopsy within 30 days post-transplant.
* Positive DSA as detected by magnetic microbeads using a Luminex® system.
* Age ≥ 18 years.
* Women of child-bearing potential (CBP) must have negative pregnancy test at screening.
* Women of CBP and men with sexual partners of CBP must agree to use a medically acceptable method of contraception throughout the study and for 3 months following discontinuation of assigned treatment.
* Subjects must be capable of understanding the purpose and risks of the study and must sign a statement of informed consent.

Exclusion Criteria:

* Recipients of multi-organ transplants.
* Recipients with previous early AMR.
* Recipients with a known hypersensitivity to C1INH, rabbit anti-thymocyte globulin, or any rabbit protein.
* History of malignancy within 3 years of enrollment (except for adequately treated basal cell or squamous cell carcinoma of the skin).
* Subjects who are positive for hepatitis C, hepatitis B surface antigen, or HIV at the time of transplant.
* Subjects who are actively taking an investigational drug.
* Subjects with a history of a psychological illness or condition that could interfere with the subject's ability to understand the requirements of the study.
* Female subjects who are pregnant or nursing.
* Subjects with hemodynamic instability, as defined by a mean arterial pressure (MAP) <60 mmHg or >110 mmHg; or requirement of vasopressors to maintain a MAP of 60 mmHg; or requirement of IV vasodilators for hypertensive emergency; or acute pulmonary edema.
* Subjects with known active infection at the time of enrollment.
* Biopsy-confirmed concurrent cellular rejection requiring polyclonal antibody therapy (i.e., all Grades other than Banff 1a and 1b will be excluded).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy will be defined as renal allograft survival 6 months following treatment for AMR. Renal allograft loss will be defined as either (1) subject death, (2) return to dialysis for greater than 30 days, or (3) re-transplantation. | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Hans Sollinger, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States